CLINICAL TRIAL: NCT04145323
Title: Novel Application of Indocyanine Green as a Biomarker to Identify Tissue Necrosis in Mastectomy Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 2019-0557; SMPH/SURGERY/SURGTRAMA (Other: UW, Madison); A539714 (Other: UW, Madison); UW19043 (Other: UW Carbone Cancer Center)
Record Dates: First submitted 2019-10-28; First posted 2019-10-30 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; Necrosis
Keywords: mastectomy; Breast reconstruction; necrosis; Indocyanine Green
MeSH Terms: conditions — Breast Neoplasms; Necrosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- ICG microangiography for necrotic tissue determination (Experimental): During flap procedure, the study area of the patient will be imaged with a white light digital camera prior to a 5 mg dose of ICG as per FDA approved protocol for use of SPY device in microangiography. Following ICG injection, the study area will undergo fluorescence imaging using the SPY system to obtain microangiography perfusion data (baseline imaging - Standard of Care). During the standard postoperative evaluation (approximately 4 hours after baseline) and 24 hours after baseline, the study area will undergo repeat digital photography and fluorescence imaging using SPY for necrosis avid detection of ICG (Research only session). This evaluation with digital photography and fluorescence imaging will continue every 24 hours for the first 3 days after surgery or one day prior to discharge(Research only session).
  Interventions: Diagnostic Test: ICG microangiography

INTERVENTIONS:
Diagnostic Test: ICG microangiography — Indocyanine Green (ICG) is a FDA approved dye which preferentially bind to exposed phospholipids in the membranes of necrotic cells, thus acting as a biomarker for necrotic tissue.

SUMMARY:
Breast reconstruction is a common procedure that can dramatically improve the quality of life and satisfaction for women who undergo mastectomy, with over 100,000 procedures performed in the U.S. in 2018. The success of this procedure, however, is limited by its complications, including mastectomy skin flap necrosis, which occurs at a rate a 10-15%. Mastectomy skin flap necrosis causes significant morbidity in patients undergoing breast reconstruction, potentially compromising results and delaying oncologic management. In addition, necrosis can lead to infection, implant loss, and need for reoperation.

Current approaches to identify mastectomy skin flap necrosis rely largely on the surgeon's assessment of skin flap color, capillary refill, temperature turgor and dermal bleeding. However, clinical assessment of necrosis is subjective and is not a reliable predictor of postoperative complications. ICG microangiography is an accepted adjunct method to aid in clinical judgment by identifying poor perfusion as a surrogate marker for tissue at risk for necrosis during reconstructive surgical procedures. However, transient alterations in blood flow seen by this method may not represent actual necrosis. Furthermore, the common practice of using vasoconstriction methods to prevent massive blood loss in plastic surgery also alters microperfusion and renders the microangiography inaccurate. There is an unmet need for reliable methods to identify mastectomy skin flap necrosis during or post breast reconstruction procedure in order to improve patient outcomes.

Recently in animal models of burn or ischemic injuries, ICG dye was shown to preferentially bind to exposed phospholipids in the membranes of necrotic cells, thus acting as a biomarker for necrotic tissue, when imaged a day after injection rather than minutes after injection, as is standard for microangiographic use of ICG. This necrosis-avid property of ICG has broad translational potential for clinical use in a variety of disease processes that result in necrosis. However, no clinical application of the necrosis-avid property of ICG has been reported yet. In this study, the investigator will test the feasibility of combining the necrosis-avid property of ICG and the SPY imaging system at University of Wisconsin hospital to obtain delayed imaging of ICG fluorescence for direct necrosis detection in breast reconstruction in mastectomy patients.

This project is an early feasibility study to establish whether ICG imaging, in a delayed fashion, can be used in mastectomy patients to aid in the detection of necrotic tissue in breast reconstruction wounds. Investigators will use the preliminary data generated from this pilot study to generate hypotheses and to power future studies.

ELIGIBILITY:
Inclusion Criteria:

* Female, age 18 years or older
* Subject undergoes mastectomy
* Subject receives intraoperative ICG during their breast reconstruction procedure
* Subject is expected to need at least 4 days of hospitalization as determined by the attending plastic surgeon on admission
* Subject understands the study procedures and can provide informed consent to participate in the study and authorization for release of relevant protected health information to the study investigator.

Exclusion Criteria:

* Subject has known contraindication to ICG injection, i.e. previous reaction to ICG (adverse event rate 1 in 42,00010)
* Subject has Iodine allergy
* Subject is pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Comparison of Necrotic tissue area determined visually by the operating surgeon vs indocyanine Green (ICG) microangiography | 24 hour post ICG injection
  Compare the risk of necrosis as determined visually by the operating surgeon at the time of mastectomy and reconstruction vs using microangiographic properties of ICG.
Time to achieve the peak fluorescent signal from necrotic tissue using ICG | up to 3 days
  Sequential fluorescence images of necrotic tissue identified by ICG fluorescence will be collected over time to identify the peak signal of fluorescence and determine correlation to time from surgery.
Percentage overlap of identified areas of necrosis determined by ICG and clinical standard of care | up to 3 days
  Compare identified areas of necrosis between ICG and clinical outcome to determine the percentage overlap of necrosis.

CONTACTS AND LOCATIONS:
Overall Officials: Angela L Gibson, MD, PhD, Principal Investigator — University of Wisconsin, Madison; Samuel O Poore, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No